CLINICAL TRIAL: NCT03328312
Title: A Randomized, Blinded, Prospective Study of the Combined Use of Low-dose Sugammadex Plus Neostigmine Administered for Reversal of Rocuronium-induced Neuromuscular Block in Obese Patients
Brief Title: Combined Use of Low-dose Sugammadex Plus Neostigmine Administered for Reversal of Rocuronium
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Breazu Caius Mihai, Assistant professor MD,PhD, Iuliu Hatieganu University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 36325348/2017
Record Dates: First submitted 2017-10-17; First posted 2017-11-01 (Actual); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Incidence of Postoperative Residual Curarization
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sugammadex (Active Comparator): For reversal of rocuronium neuromuscular- block we will use Sugammadex
  Interventions: Drug: Sugammadex
- neostigmine+atropine (Placebo Comparator): For reversal of rocuronium neuromuscular- block we will use Neostigmine (Miostin®; Stigmosan®) 0.05 mg/kg and atropine 1 mg/ dose.
  Interventions: Drug: neostigmine+atropine
- neostigmine+atropine+sugammadex (Experimental): For reversal of rocuronium neuromuscular- block we will use Neostigmine (Miostin®; Stigmosan®) 0.025 mg/kg and atropine 0.5 mg/dose followed within 3 min by Sugammadex 1 mg/kg.
  Interventions: Drug: neostigmine+atropine+sugammadex

INTERVENTIONS:
Drug: Sugammadex — Time period from administration of the reversal agent to recovery of TOFR >0.9
  Arms: Sugammadex
Drug: neostigmine+atropine — Number and time of bradycardic episodes (HR<60 bpm) as well as that of tachycardic episodes (HR>100 bpm) before tracheal extubation
  Arms: neostigmine+atropine
Drug: neostigmine+atropine+sugammadex — 4. Time of extubation
  Arms: neostigmine+atropine+sugammadex

SUMMARY:
Reversal of rocuronium-induced neuromuscular block by the combination of low-doses of neostigmine plus sugammadex decreases the cost of anesthetic medications, while maintaining efficacy of reversal in obese patients.

DETAILED DESCRIPTION:
Background Neuromuscular paralysis is a frequent requirement to facilitate airway management and surgery. Patients receiving neuromuscular blocking agents (NMBAs) are at risk of residual neuromuscular blockade (RNMB) that can lead to postoperative cardio-pulmonary complications, and may increase postoperative morbidity and mortality.1-2 NMBAs can be antagonized with the cholinesterase inhibitor neostigmine; however, this agent has several undesirable side effects because of its parasympathetic stimulation.3 Thus, muscarinic receptor antagonists, such as atropine, are used along with cholinesterase inhibitors; however, these drugs also have their own set of adverse effects. Despite its relatively slow onset of action and inability to antagonize profound blockade, neostigmine is still used frequently for reversal of rocuronium-induced neuromuscular blockade because of its low cost. Sugammadex is a selective relaxant biding agent, developed to encapsulate the steroidal NMBAs, and proved to be extremely effective for the reversal of either shallow (dose of 2 mg/kg), deep (dose of 4 mg/kg), or even profound (dose of 16 mg/kg) neuromuscular blockade. However, routine use of sugammadex is limited by its relatively high cost compared with neostigmine.

The purpose of the study is to investigate drug costs and adverse effects of low-dose neostigmine (0.025 mg/kg) plus low-dose sugammadex (1 mg/kg) for reversal of rocuronium-induced neuromuscular block, and compare efficacy of antagonism and costs of this combination therapy with the current standard therapies: full-dose sugammadex (2 mg/kg) and full-dose neostigmine (0.05 mg/kg) plus atropine.

Randomization and blinding On randomization, each patient will be allocated by a unique identifying number into study groups "A", "B", or "C". The allocation of a patient to the specific group will be only known by the research assistant. The participating anaesthetists as well as the research staff who collect patient data will remain blinded until after the completion of the study.

For reversal of rocuronium neuromuscular- block we used:

* Group A - Sugammadex (Bridion®) 2 mg/kg,
* Group B - Neostigmine (Miostin®; Stigmosan®) 0.05 mg/kg and atropine 1 mg/ dose.
* Group C - Neostigmine (Miostin®; Stigmosan®) 0.025 mg/kg and atropine 0.5 mg/dose followed within 3 min by Sugammadex 1 mg/kg.

Monitoring the neuromuscular blockade After induction of anesthesia and before administration of rocuronium, monitoring of neuromuscular blockade at the adductor pollicis muscle is initiated using acceleromyography (TOF-Watch SX, Organon, Dublin, Ireland). After degreasing the skin, two surface electrodes are placed above the ulnar nerve near the wrist. After induction of general anesthesia, 50-Hz tetanic stimulation is applied for 5 sec and followed after 1 min by train-of-four (TOF) stimulation every 15 sec. If the response to TOF is stable, calibration and supramaximal stimulation are ensured by built-in calibration function (CAL2). After at least 2 min of a stable baseline documentation of the response to TOF, rocuronium is administered.

At the end of surgery, inhalational agent (sevoflurane) will be discontinued. Once the end-tidal concentration of sevoflurane reaches 0.4-0.6%, the previously randomized reversal study drug will be administrated at shallow neuromuscular block (TOF count of 2). The primary efficacy variable is the incidence of residual neuromuscular block (defined as TOFR <0.90) measured at least 15 min. after the administration of the reversal agent. In case of residual block, a rescue dose of 2 mg/kg sugammadex will be administrated before tracheal extubation. Extubation is performed once patient is deemed fully recovered (TOFR = 1.0)

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective abdominal surgery
* 16-65 years of age
* BMI 30-39.9 ( obese class I-II)
* American Society of Anesthesiologists (ASA) physical status II.
* Surgery scheduled for general anesthesia and tracheal intubation and planned extubation at the end of surgery
* Surgical procedures with an anticipated length of at least 60 min.

Exclusion Criteria:

* Emergency surgery

  * Patients unable to consent to study participation
  * Patients expected to be maintained on mechanical ventilation postoperatively
  * Contraindication to any of the study drugs
  * Patients with existing neuromuscular disease
  * Acute or chronic renal failure (GFR-EPI <30 mL/min/1.73 m2)
  * Acute/chronic liver disease (Child-Pugh Score >1)
  * Hyperkalemia (> 5.3 mmol/l)
  * Pregnancy
  * History of stroke or ongoing paresis
  * Glaucoma
  * Breast feeding
  * Sepsis

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative residual curarization (PORC) | 24 hours
  Incidence of postoperative residual curarization (PORC) (defined as a train-of-four ratio, TOFR <0.9) measured 15 min after administration of the reversal agent.

SECONDARY OUTCOMES:
Time | 24 hours
  1. Time period from administration of the reversal agent until recovery of TOFR to >0.90
Bradycardia | 24 hours
  2. Number of bradycardic episodes (HR <60 bpm).
Residual blockade | 24 hours
  3. Incidence of clinical symptoms potentially associated with residual neuromuscular blockade (diplopia, difficulty swallowing, feeling of general weakness)

CONTACTS AND LOCATIONS:
Overall Officials: Caius Breazu, Md,PhD, Principal Investigator — Iuliu Hatieganu University of medicine and pharmacy cluj-Napoca

IPD SHARING:
Plan to Share IPD: Undecided